CLINICAL TRIAL: NCT03231319
Title: Comparison of Different Neural Blockade Techniques in Postoperative Analgesia After Total Hip Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CF17089A
Record Dates: First submitted 2017-06-22; First posted 2017-07-27 (Actual); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Analgesia, Patient-Controlled

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- fascia iliaca compartment block+ IV-PCA (Active Comparator)
  Interventions: Procedure: Fascia iliaca compartment block with IV-PCA
- femoral nerve and lateral femoral cutaneous nerve block+IV PCA (Active Comparator)
  Interventions: Procedure: Femoral nerve block and lateral femoral cutaneous nerve with IV-PCA
- IV PCA only (Placebo Comparator)
  Interventions: Procedure: IV-PCA

INTERVENTIONS:
Procedure: Fascia iliaca compartment block with IV-PCA — 1. Fascia iliaca compartment block: The injection was performed under ultrasound guidance. Surface landmark is identified on the line between anterior superior iliac spine and pubic tubercle. The injection site is at the medial one-third of the line. The needle is threaded medial to lateral and standardization of local anesthetic deposit is in the fascia plane between fascia iliaca and iliacus muscle. Anesthetic regimen: 2% xylocaine 15mL + 0.5% bupivacaine 15mL.
  Arms: fascia iliaca compartment block+ IV-PCA
Procedure: Femoral nerve block and lateral femoral cutaneous nerve with IV-PCA — 1. Femoral nerve block: The injection was performed under ultrasound guidance. Femoral nerve was identified in the femoral neurovascular bundle below or around inguinal ligament. The needle is threaded with lateral to medial approach. Local anesthetics will be deposited around the femoral nerve, the standardization of protocol is that femoral nerve should be lifted off from iliacus muscle. Anesthetic regimen: 2% xylocaine 10mL + 0.5% bupivacaine 10mL.
  2. Lateral femoral cutaneous nerve block: The injection was performed under ultrasound guidance. Lateral femoral cutaneous nerve was identified in the fascia plane between sartorius muscle and tensor fascia lata muscle. Anesthetic regimen: 2% xylocaine 5mL + 0.5% bupivacaine 5mL
  Arms: femoral nerve and lateral femoral cutaneous nerve block+IV PCA
Procedure: IV-PCA — IV-PCA was programmed and provided to the patient for optimize pain control
  Arms: IV PCA only

SUMMARY:
To compare the different analgesic protocols for patients receiving total hip arthroplasty(THA). Patients will divided into 3 groups, which are 1. fascia iliaca compartment block with IV-PCA(patient controlled analgesia), 2. femoral nerve and lateral femoral cutaneous nerve block with IV-PCA, 3. IV-PCA only.

DETAILED DESCRIPTION:
90 patients will be enrolled and randomized to the 3 different groups.

1. Inclusion criteria:

   Patient undergoing THA: 20-75 years old, ASA I-III, general anesthesia with intubation, fentanyl IV PCA.
2. Exclusion criteria Alcohol/substance abuse Rheumatoid arthritis Severe coagulation disorder(PLT<80000 or INR > 1.5) Peripheral neuropathy Allergy to opioids or local anesthetics BMI>35
3. The outcome followers are blinded to the intervention provided.
4. Outcome parameters:

   1. Opioid consumption of IV PCA in first 24 hrs.
   2. NSAID consumption
   3. NRS of pain, the timings of follow-up should be: pre-block, 30

      mins post-block, 60 mins post-block, 2 hours post-block, 24hours post-block
   4. sensory block in FN, Obturator Nerve and LFCN
   5. First request of supplemental IV analgesia

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III, general anesthesia with intubation.
* fentanyl IV PCA

Exclusion Criteria:

* Alcohol/substance abuse
* Rheumatoid arthritis
* Severe coagulation disorder(PLT<80000 or INR > 1.5)
* Peripheral neuropathy
* Allergy to opioids or local anesthetics
* BMI>35

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-07-27 (Estimated); Primary Completion 2018-04-19 (Estimated); Study Completion 2018-04-19 (Estimated)

PRIMARY OUTCOMES:
Temporal changes of Pain score | 1. Pre-intervention(which is the time when operation was done and the patient arrive postoperative care unit.) 2. 30 minutes after intervention, 3. 60 minutes after intervention, 4. 120 minutes after intervention, 5. 24 hours after intervention.
  Pain score by numerical rating scale from pre-intervention to 24 hours after intervention(the effect of neural blockade seldom lasts more than 24 hours)

SECONDARY OUTCOMES:
Opioid consumptions | postoperatively 24 hours
  Including IV-PCA and other analgesics
Sensory block in femoral nerve, obturator nerve and lateral femoral cutaneous nerve area | 1 hour post-intervention
NSAID consumptions | 24 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Ting Chang, M.D., Study Chair — Taichung Veterans General Hospital
Locations (2):
- Taiwan (2):
  - Taichung Veterans General Hospital, Taichung
  - Dept. of Anesthesiology, Taichung Veterans General Hospital, Taichung

REFERENCES:
- [Background] 1. Hadzic's peripheral nerve blocks and anatomy for ultrasound-guidedregional anesthesia, 2012. Chapter.35, 36. 2. K.H. Thymo, O. Mathiesen, J.B. Dahl, et al. Lateral femoral cutaneous nerve block after total hip arthroplasty: a randomized trial. Acta Anaesthesiologica Scandinavica 60(2016) 1297-1305. 3. Shoji Nishio, Shigeo Fukunishi, Miura Juichi et al. Comparison of continuous femoral nerve block, caudal epidural block, and intravenous patient-controlled analgesia in pain control after total hip arthroplasty: a prospective randomized study. Orthopedic Reviews 2014; 6; 5138. 4. Bin Yu, Miao He, Guang-Yu Cai et al. Ultrasound-guided continuous femoral nerve block vs continuous fascia iliaca compartment block for hip replacement in the elderly. Medicine (2016) 95:42 5. Guay J, Parker MJ, Gajendragadkar PR, et al. Anaesthesia for hip fracture surgery in adults. Cochrane Database of Systemic Reviews 2016, issue 2, Art. No:CD000521. 6. K.H. Thybo, Harald Schmidt and Daniel Hagi-Pederson. Effect of lateral femoral cutaneous nerve block on pain after total hip arthroplasty: a randomized , blinded, placebo-controlled trail. BMC anesthesiology (2016) 16:21. 7. John Dolan, Anne Williams, Eileen Murney, et al. Ultrasound guided fascial iliaca block: a comparison with loss of resistance technique. Reg Anesth Pain Med 2008; 33: 526-31 8. Ali N. Shariat, Admir Hadzic, Daquan Xu, et al. Fascia iliaca block for analgesia after hip arthroplasty: a randomized double-blinded, placebo-controlled trial. Reg Anesth Pain Med 2013;38:201-205